CLINICAL TRIAL: NCT04792658
Title: Impact of Long Term of Benzodiazepine Use on Psychiatric Manifestation in Neuropsychiatric Disease
Brief Title: Impact of Long Term of Benzodiazepine Use on Psychiatric Manifestation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer, resarcher OF Neurology and Psychiatry department, Assiut University
Other Study IDs: long term of benzodiazepine
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Psychiatric Disorder; Benzodiazepine-Related Disorders
Keywords: psychiatric; benzodiazepine
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Detailed interview with personal demographic data — , such as age, sex, education, history of occupation, past medical history, family history, medical, neurological, and psychiatric disorders.
Behavioral: Intelligence assessment using the Arabic version of the Wechsler Adult Intelligence Scale (WAIS) — the test consists of six verbal subtests and five performance subtests. It used in measure Intelligence
Behavioral: The Arabic version of the Structured Interview for the Five-Factor Personality Model (SIFFM) — it depend on a model of general language personality descriptors that based on theory suggests five broad dimensions to describe human personality
Behavioral: the Hamilton Depression Rating Scale — it used for evaluation depression severity. It is 17 items and each item's score (0-4). with a total score range of 0-54
Behavioral: The Hamilton Anxiety Rating Scale — it used for evaluation the severity of anxiety. The scale consists of 14 items and each item is scored on a scale from 0 to 4 , with a total score range of 0-56
Behavioral: The Minnesota Multiphasic Personality Inventory-2 (MMPI-2) — It used to evaluate range of symptoms of psychopathology and personality traits that are maladaptive. It has 10 clinical scales subscales included the following: 1, hypochondriasis (Hs); 2, depression (D); 3, hysteria (Hy); 4, psychopathic deviation (Pd); 5, masculinity-femininity (Mf); 6, paranoia (Pa); 7, psychophrenia (Pt); 8, schizophrenia (Sc); 9, hypomania (Ma); 10, social introversion (Ma); (Si). More than 65 responses were considered symptomatic

SUMMARY:
Benzodiazepines are usually a secondary drug of abuse-used mainly to augment the high received from another drug or to offset the adverse effects of other drugs. Few cases of addiction arise from legitimate use of benzodiazepines. Pharmacologic dependence, a predictable and natural adaptation of a body system long accustomed to the presence of a drug, may occur in patients taking therapeutic doses of benzodiazepines. However, this dependence, which generally manifests itself in withdrawal symptoms upon the abrupt discontinuation of the medication, may be controlled and ended through dose tapering, medication switching, and/or medication augmentation. Due to the chronic nature of anxiety, long-term low-dose benzodiazepine treatment may be necessary for some patients; this continuation of treatment should not be considered abuse or addiction.

previous study reported that The results of the study are important in that they corroborate the mounting evidence that a range of neuropsychological functions are impaired as a result of long-term benzodiazepine use, and that these are likely to persist even following withdrawal. The findings highlight the residual neurocognitive compromise associated with long-term benzodiazepine therapy as well as the important clinical implications of these results.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 years to 50 years
* No history of neurological or medical illness

Exclusion Criteria:

* intelligence score more than 80

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participants who have use benzodiazepine more than 1 year and attend in outpatient clinic in Neuropsychiatric department will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
measure the prevalence of DSM 5 psychiatric disorders associated with long term of benzodiazepine use | through study completion, an average of 1 year
measure of risk factor of DSM 5 psychiatric disorders associated with long term of benzodiazepine use | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shinfuku M, Kishimoto T, Uchida H, Suzuki T, Mimura M, Kikuchi T. Effectiveness and safety of long-term benzodiazepine use in anxiety disorders: a systematic review and meta-analysis. Int Clin Psychopharmacol. 2019 Sep;34(5):211-221. doi: 10.1097/YIC.0000000000000276. PMID 31274696
- [Result] O'brien CP. Benzodiazepine use, abuse, and dependence. J Clin Psychiatry. 2005;66 Suppl 2:28-33. PMID 15762817
- [Result] Crowe SF, Stranks EK. The Residual Medium and Long-term Cognitive Effects of Benzodiazepine Use: An Updated Meta-analysis. Arch Clin Neuropsychol. 2018 Nov 1;33(7):901-911. doi: 10.1093/arclin/acx120. PMID 29244060